CLINICAL TRIAL: NCT01071720
Title: Clinical Study to Assess the Effect of Food on the Pharmacokinetic Characteristics of CKD-501 in Healthy Subjects
Brief Title: The Effect of Food on the Pharmacokinetic Characteristics of CKD-501
Acronym: CKD-501 FDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Soo-Yeon Kim/CRA, Chong Kun Dang Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CKD-19HPS09L
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-501 1mg (fed-fasted group) (Other): CKD-501 1mg should be administered following a high-fat, high-caloric diet(fed condition) in one period and on an empty stomach(fasting condition) in the other period.
  Interventions: Drug: CKD-501 1mg
- CKD-501 1mg (fasted-fed group) (Other): CKD-501 1mg should be administered on an empty stomach(fasting condition) in one period and following a high-fat, high-caloric diet(fed condition) in the other period.
  Interventions: Drug: CKD-501 1mg

INTERVENTIONS:
Drug: CKD-501 1mg — This study is randomized, balanced, single-dose, two treatment (fed versus fasting), two-period, two sequence crossover design to assess the effects of food on pharmacokinetics profile.

SUMMARY:
The purpose of this study is to assess the effect of food on the pharmacokinetic characteristics of CKD-501 in healthy subject.

And, secondarily, pharmacokinetic characteristics of the main metabolites will be identified.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose (CKD-501 1mg), two treatment(fed vs. fasting), two-period, two sequence crossover.

Every time before and after each medication, PK parameters and safety of CKD-501 1mg is performed using a blood sample and conducting some tests respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 aged in healthy adults
* Weight more than 45kg, IBW 20% within the range
* Agreement with written informed consent

Exclusion Criteria:

* Subject has symptoms of acute disease within 28 days of starting administration of investigational drug
* Subject with known for history(such as inflammatory gastrointestinal disease, gastric or duodenal ulcer, liver diseases and so on) with affect the ADME of drug
* Clinically significant, active gastrointestinal system, cardiovascular system, pulmonary system, renal system, endocrine system, blood system, digestive system, central nervous system, mental disease or malignancy disease
* Inadequate subject by medical examination(medical history, physical examination, ECG, laboratory test) within 28 days of starting administration of investigational drug
* Inadequate result of laboratory test

  * AST(SGOT) or ALT(SGPT) > 1.25 x upper limit of normal range
  * Total bilirubin > 1.5 x upper limit of normal range
* Clinically significant allergic disease(Except for mild allergic rhinitis seems to be not need for medication)
* Subject with known for hypersensitivity reactions to glitazone
* Previously participated in other trial within 60 days
* Treatment with dug-medicated induction/inhibition metabolic enzyme such as barbiturates within 1 month or with may affect the clinical trial within 10 days
* Subject takes an abnormal meal which affect the ADME of drug
* Not able to taking the institutional standard meal
* Previously make whole blood donation within 60 days or component blood donation within 20 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 30 g/day) or during clinical trials can not be drunk or severe heavy smoker (cigarette > 10 cigarettes per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result
* Subject who not practice contraception during clinical trial or pregnant women(including positive pregnancy test) or nursing mothers

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of CKD-501 1mg (fed vs. fasting) | 0-48 hrs

SECONDARY OUTCOMES:
To evaluate the safety of CKD-501 1mg from vital signs, physical exam, ECG, laboratory test, adverse event and so on | Throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, Ph.D., Principal Investigator — Korea University Anam Hospital